CLINICAL TRIAL: NCT00883831
Title: Acupuncture for Symptomatic Care of Hemodialysis Patients: a Case-series
Brief Title: The Effectiveness and the Safety of Acupuncture for Symptomatic Care of Hemodialysis Patients: A Case-series
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Korea Institute of Oriental Medicine (Other Government)
Responsible Party: Korea Institute of Oriental Medicine, Korea Institute of Oriental Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KI0904
Record Dates: First submitted 2009-04-17; First posted 2009-04-20 (Estimated); Last update posted 2010-01-25 (Estimated); Status verified 2009-04

CONDITIONS: Hemodialysis; End Stage Renal Disease
Keywords: Acupuncture; Hemodialysis; Symptom; end stage renal disease; chronic kidney disease; supportive care
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Individualized manual acupuncture (Experimental)
  Interventions: Procedure: Individualized manual acupuncture

INTERVENTIONS:
Procedure: Individualized manual acupuncture — Acupuncture treatment will be provided according to traditional korean medicine (TKM) theory which focuses on patient's individual symptoms and conditions. 10-12 needles will be inserted into acupuncture point on the body except one arm where arteriovenous fistula is located for hemodialysis access. Needle retention time will be 30 minutes with intermittent manual stimulation to elicit de-qi sensation. Biweekly treatment will be conducted at non-dialysis access day or before hemodialysis at dialysis-access day for 6 weeks.

SUMMARY:
Purpose:

Hemodialysis-dependent patients with an end-stage renal disease (ESRD) suffer from a number of distressing symptoms, such as pain, poor mental health, fatigue, sleep disturbance and pruritus. These negatively influence health-related quality of life in ESRD patients, and some of them result in increased mortality and hospitalization. Acupuncture is a widely employed treatment on several chronic disease or condition. Adjunctive use of acupuncture with conventional treatment could be a possible therapeutic option to establish an optimal care for ESRD patients who experiences co-morbid conditions or complications of hemodialysis. Due to its non-pharmacologic feature, the effects of acupuncture without involving altered pharmacokinetics and drug-interactions in hemodialysis patients, might be another strong point compared to other pharmacological interventions. However, little information is available for the effects and the safety of acupuncture for symptomatic care of hemodialysis patients.

Thus, the investigators propose whether acupuncture could be a effective and safe therapeutic modality for a number of patient-reported symptoms in hemodialysis-dependent patients with ESRD.

DETAILED DESCRIPTION:
This trial is a case-series, with a nested-qualitative study at the end of follow-up. Acupuncture treatment will be provided biweekly for 6 weeks, namely total 12 sessions, and follow-up period will be 4 weeks after the end of treatment. Changes of symptoms, quality of life and occured adverse events will be assessed during study procedure. Patients who agreed joining qualitative research will be interviewed about their experiences of acupuncture in detail.

ELIGIBILITY:
Inclusion Criteria:

* over 19 years old
* started hemodialysis at least 3 months ago
* receiving hemodialysis 3 times a week regularly
* equilibrated Kt/V ≥ 1.2
* willingness to participate in this study

Exclusion Criteria:

* acute/chronic liver disease
* events of life-threatening cardiovascular disease within 6 months
* events of life-threatening neurological disorder within 6 months
* current/past history of neoplasm
* hemorrhagic disorders
* drug abuse/alcoholism
* other infectious disease including active tuberculosis
* history of the use of acupuncture, moxibustion or herbs within 1 month

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2009-04; Primary Completion 2009-12 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Measure Your Medical Outcome Profile2 (MYMOP) | Evaluated at baseline, post-treatment, and 4 weeks after post-treatment (total 3 times)

SECONDARY OUTCOMES:
Kidney Disease Quality of Life-SF V1.3 (KDQOL-SF V 1.3) questionnaire | Evaluated at baseline, post-treatment, and 4 weeks after post-treatment (total 3 times)

CONTACTS AND LOCATIONS:
Overall Officials: Sun Mi Choi, PhD, Principal Investigator — Korea Institute of Oriental Medicine
Locations (1):
- Doonsan Oriental Hospital of Daejeon University, Daejeon, South Korea

REFERENCES:
- [Derived] Kim KH, Kim TH, Kang JW, Sul JU, Lee MS, Kim JI, Shin MS, Jung SY, Kim AR, Kang KW, Choi SM. Acupuncture for symptom management in hemodialysis patients: a prospective, observational pilot study. J Altern Complement Med. 2011 Aug;17(8):741-8. doi: 10.1089/acm.2010.0206. Epub 2011 Jul 1. PMID 21721925